CLINICAL TRIAL: NCT06608160
Title: 68Ga-grazytracer PET/CT Assists in Diagnosing Pseudoprogression Following Immunotherapy in Lung Cancer: a Prospective, Observational Study.
Brief Title: 68Ga-grazytracer PET Assists in Diagnosing Pseudoprogression Following Immunotherapy in Lung Cancer.
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-350
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: PET / CT; Lung Carcinoma; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, there are limited methods available in clinical practice to distinguish pseudoprogression after immunotherapy. Most patients rely on follow-up observations to monitor the disease, which does not meet clinical needs. 68Ga-grazytracer is a novel imaging agent targeting granzyme B. By detecting the concentration of granzyme B, it reflects the localization of cytotoxic T cells in the tumor region and their potential ability to kill tumor cells. This study aims to leverage the simplicity, non-invasiveness, visualization, and semi-quantitative advantages of 68Ga-grazytracer PET imaging to evaluate its effectiveness and feasibility in diagnosing pseudoprogression.

ELIGIBILITY:
Inclusion Criteria:

1. Lung cancer patients who develope lesion enlargement and/or new lesions after treatment with immune checkpoint inhibitors;
2. Pseudoprogression cannot be ruled out in clinical practice;
3. Lung cancer confirmed by pathology or cytology, regardless of pathological type;
4. Fully-informed written consent obtained from patients;
5. Patient ability to comply with protocol requirements;
6. Age 18-75 years;
7. Life expectancy of at least 6 months.

Exclusion Criteria:

1. Patients with serious diseases that the investigator deems unsuitable for participation in the clinical study. Such as severe cardiopulmonary insufficiency, severe bone marrow suppression, severe hepatic or renal insufficiency, etc;
2. Intestinal perforation, complete intestinal obstruction;
3. Active phase of hepatitis B；
4. Pregnant women and women who are potentially pregnant, as well as nursing mothers;
5. Patients with poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are enrolled from Department of Respiratory and Critical Care Medicine, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine in China.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance 1 | Follow-up for 4-8 weeks, not exceeding 12 weeks.
  Sensitivity and specificity of 68Ga-grazytracer PET in diagnosing pseudoprogression

SECONDARY OUTCOMES:
Diagnostic performance 2 | Follow-up for 4-8 weeks, not exceeding 12 weeks.
  Investigating the optimal uptake value for 68Ga-grazytracer PET/CT imaging in diagnosing pseudoprogression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China